CLINICAL TRIAL: NCT05561569
Title: Randomized Trial Comparing Air Versus Gas Tamponade in Primary Retinal Detachment
Brief Title: Air Versus Gas Tamponade in Primary Retinal Detachment
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Benha University (Other)
Responsible Party: Principal Investigator, Ahmed Abdelshafy, Assistant professor of Ophthalmology, Benha University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Rc.11-2022
Record Dates: First submitted 2022-09-26; First posted 2022-09-30 (Actual); Last update posted 2022-09-30 (Actual); Status verified 2022-09

CONDITIONS: Retinal Detachment; Proliferative Vitreoretinopathy
Keywords: Vitrectomy; Retinal detachment
MeSH Terms: conditions — Retinal Detachment; Vitreoretinopathy, Proliferative

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Air tamponade group (Active Comparator): Cases with primary upper retinal detachment that will be treated with air tamponade.
  Interventions: Procedure: Pars plana vitrectomy
- Non expansile gas tamponade group (Active Comparator): Cases with primary upper retinal detachment that will be treated with sulfur-hexafluoride 6 (SF-6) gas tamponade.
  Interventions: Procedure: Pars plana vitrectomy

INTERVENTIONS:
Procedure: Pars plana vitrectomy — 23 gauge pars plana vitrectomy for managing primary retinal detachment.

SUMMARY:
Management of primary retinal detachment due to upper retinal break is one of controversial situation that may face ophthalmologists in vitreoretinal subspecialty.

DETAILED DESCRIPTION:
There is no single surgical plan for management of primary retinal detachment due to upper retinal break, some surgeons prefer scleral buckling over vitrectomy in cases with no traction over the retinal break, others prefer to perform primary pars-plana vitrectomy with either air or gas tamponade.

In this study we aim to compare the results of air and non-expansile gas tamponade in cases with upper retinal detachment with grade a or b proliferative vitreoretinopathy.

ELIGIBILITY:
Inclusion Criteria:

* primary rhegmatogenous retinal detachment with upper break with proliferative vitreoretinopathy from grade a to b.

Exclusion Criteria:

* cases with combined tractional retinal detachment.
* cases with recurrent retinal detachment.
* cases that are eligible for scleral buckling that have no traction on retinal break.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2022-09-26 (Actual); Primary Completion 2023-06-01 (Estimated); Study Completion 2023-07-01 (Estimated)

PRIMARY OUTCOMES:
Improvement in visual acuity | Change from baseline visual acuity at 6th month.
  Visual acuity changes measured by snellen chart and converted to LogMar units.

SECONDARY OUTCOMES:
Changes in metamorphopsia | Change from baseline metamorphopsia at 6th month.
  Changes in metamorphopsia after surgery assessed by M-chart that is specially designed to subjectively assess metamorphopsia, each 1 millimeter deviation from reference line is considered significant deviation.

OTHER OUTCOMES:
Recurrence of retinal detachment | Incidence of recurrent retinal detachment at 6th month.
  Incidence of recurrent retinal detachment in each group assessed by indirect fundus ophthalmoscope.

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed A Abdelshafy, MD, Principal Investigator — Benha University
Locations (1):
- Ahmed Abdelshafy, Banhā, QA, Egypt

IPD SHARING:
Plan to Share IPD: No